CLINICAL TRIAL: NCT02682069
Title: A Prospective, Single-blind Evaluation of the Positive Predictive Value (PPV) of the MolecuLight i:X(TM) Imaging Device to Predict the Presence of Bacteria in Chronic Wounds
Brief Title: Positive Predictive Value of the MolecuLight i:X Imaging Device to Predict the Presence of Bacteria in Chronic Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MolecuLight Inc. (Industry)
Collaborators: Southwest Regional Wound Care Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: 16-001
Record Dates: First submitted 2016-02-08; First posted 2016-02-15 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Wounds
Keywords: Diabetic foot ulcer; venous leg ulcer; fluorescence imaging; wound imaging
MeSH Terms: conditions — Wounds and Injuries; Diabetic Foot; Varicose Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- All patients (Experimental): There is one arm to this study and all patients will undergo the same procedures. The test of this technology is on a per wound basis where bacteria will fluoresce red and samples will be obtained from the discrete red locations. Microbiology results indicating the presence or absence of bacteria will be correlated to the fluorescence signal in the fluorescent images.
  Interventions: Device: MolecuLight i:X Imaging Device

INTERVENTIONS:
Device: MolecuLight i:X Imaging Device — The intended use of the device is to assist clinicians during care and management of patients with chronic wounds by screening for the presence of potentially harmful bacteria levels. The device will be used as part of the current clinical wound assessment process which may include examination for characteristic signs and symptoms of infection. The device can capture and document either an image or video of the chronic wound where the presence of florescent bacteria appears under violet light illumination. This information can be used to guide a clinician to inspect, sample, debride or further evaluate areas within or around a wound where fluorescent bacteria are present.

SUMMARY:
This is a non-randomized evaluation for which 50 patients will be imaged at the Southwest Regional Wound Care Center, Lubbock, Texas, who present with a chronic wound and are receiving standard treatment. The MolecuLight i:X Imaging Device will be used as an adjunctive tool in the assessment of the wound and will be used to guide the targeted sampling of a wound (punch biopsy method).

DETAILED DESCRIPTION:
MolecuLight Inc. (Toronto, Canada) has recently introduced to the Canadian market an innovative imaging device, the MolecuLight i:X™ Imaging Device, that offers real-time detection of important biological and molecular information of a chronic wound, and could have significant impact on improving conventional wound care and management. The MolecuLight i:X Imaging Device is intended to assist clinicians during care and management of patients with chronic wounds by screening for the presence of potentially harmful bacteria levels. The device can capture and document either an image or video of the chronic wound where the presence of fluorescent bacteria appears under violet light illumination. This information can be used to guide a clinician to inspect, sample, debride or further evaluate areas within or around a wound where fluorescent bacteria are present. Though the MolecuLight i:X Imaging Device has been shown to be effective in controlled settings, this study is deploying the device in a larger population and evaluating the ability of the MolecuLight i:X device to positively predict the presence of bacteria in chronic wounds.

The overall objective of this work is to evaluate the MolecuLight i:X Imaging Device in screening of chronic wounds for the presence of bacteria. The device is intended to guide the clinician to inspect, sample, debride or further evaluate areas within or around a wound where fluorescent bacteria are present.

All imaging will be performed with the MolecuLight i:X Imaging Device at an appropriate distance from the wound of interest (8 - 12 cm), which is indicated by the range finder LED. Illumination is provided by two violet (405 nm) LEDs that produce a bright, but clinically safe, uniform illumination. Fluorescence imaging is performed on the camera in real-time while the device is in fluorescence mode and the room lights are turned off. If room ambient light cannot be eliminated to an acceptable level (indicated by the ambient light sensor), the MolecuLight drape must be used to achieve a dark environment. A standard measurement sticker will be placed adjacent to the wound within the field of view to act as a reference for size.

All microbiological analysis will be performed as per standard practice at each local clinic. Tissue samples will be analyzed for culture and sensitivity, yielding the species of bacteria present in the sample (if any), the susceptibility to various antibiotics and a measure of the bacterial load.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients presenting with chronic wound of the lower limb (e.g. diabetic foot ulcer, venous leg ulcer, other acceptable aetiology)
2. 18 years or older

Exclusion Criteria:

1. Treatment with an investigational drug within 1 month before study enrolment
2. Use of systemic (oral or intravenous) antibiotics
3. Inability to consent
4. Any contra-indication to routine wound care and/or monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02; Primary Completion 2017-01-05 (Actual); Study Completion 2017-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Wolcott, MD, Principal Investigator — Southwest Regional Wound Care Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rennie MY, Lindvere-Teene L, Tapang K, Linden R. Point-of-care fluorescence imaging predicts the presence of pathogenic bacteria in wounds: a clinical study. J Wound Care. 2017 Aug 2;26(8):452-460. doi: 10.12968/jowc.2017.26.8.452. PMID 28795890

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: There is one arm to this study and all patients will undergo the same procedures.The test of this technology is on a per wound basis where bacteria will fluoresce red and samples will be obtained from the discrete red locations.Microbiology results indicating the presence or absence of bacteria will be correlated to the fluorescence signal in the fluorescent images.
Period: Overall Study
Arm/Group | All Patients
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Patients: There is one arm to this study and all patients will undergo the same procedures. The test of this technology is on a per wound basis where bacteria will fluoresce red and samples will be obtained from the discrete red locations. Microbiology results indicating the presence or absence of bacteria will be correlated to the fluorescence signal in the fluorescent images.MolecuLight i:X Imaging Device: The intended use of the device is to assist clinicians during care and management of patients with chronic wounds by screening for the presence of potentially harmful bacteria levels. The device will be used as part of the current clinical wound assessment process which may include examination for characteristic signs and symptoms of infection. The device can capture and document either an image or video of the chronic wound where the presence of florescent bacteria appears under violet light illumination.
Arm/Group | All Patients
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 24
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Positive Predictive Value (PPV) - Ability of Fluorescence Imaging With the MolecuLight i:X to Predict Presence of Bacterial Loads of 104 CFU/g and Greater
Description: PPV reflects the probability that a region of red fluorescence within or around a wound will contain bacteria. Meaning the number cases where qPCR analysis of wound tissue biopsies from red fluorescent region showed to have pathogen load ≥ 104 CFU/g divided by the total number of cases where red florescence was observed in the wound multiplied by 100,
Time Frame: Baseline
Measure: Number; unit: Percentage of PPV
Arm/Group | All Patients
Number analyzed (Participants) | 30
Percentage of PPV | 100

ADVERSE EVENTS:
Groups:
- All Patients (Imaging/no Intervention): There is only one group in this study, the imaging/no intervention group. These patients will meet all enrollment criteria and bacterial (red or cyan) fluorescence will be visualized within or around their wound with the MolecuLight i:X imaging device. A targeted curettage sample will be taken from the site of fluorescence and sent for microbiological analysis. There will be no intervention or followup.
Arm/Group | All Patients (Imaging/no Intervention)
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No